CLINICAL TRIAL: NCT06354855
Title: "Which Type of Exercise is More Effective in Chronic Constipation? (Randomized Controlled Study)"
Brief Title: "Which Type of Exercise is More Effective in Chronic Constipation?
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Fatma Erdeo, doctor, phd, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEU-FTR-FE-04
Record Dates: First submitted 2024-02-28; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Chronic Constipation

STUDY DESIGN:
Intervention Model Description: Two groups with a conventional therapy control group
Who Masked: Outcomes Assessor
Masking Description: The assignment of people to groups will be done by a statistician, apart from the research using a computer program. Randomization will be determined by entering the total number of cases through the program whose URL address is https://www.randomizer.org.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group is doing breathing exercises while watching videos (Active Comparator): Abdominal breathing exercise group .The group, which receives abdominal breathing exercise training, will perform video-assisted breathing exercises for 30 minutes a day.
  Interventions: Other: Group is doing breathing exercises while watching videos
- Medium pace walking group (Active Comparator): Medium pace walking group .Control group will walk at a moderate pace for 30 minutes daily.
  Interventions: Other: Medium pace walking group

INTERVENTIONS:
Other: Group is doing breathing exercises while watching videos — Group is doing breathing exercises while watching videos: A video consisting of 30-minute exercises will be shot for these patients. And each patient will be asked to do the breathing exercise for 30 minutes by watching this video.
  Arms: Group is doing breathing exercises while watching videos
Other: Medium pace walking group — Medium pace walking group: 30 minutes daily. Walking at a moderate pace is required. Physical activity levels will be monitored with the ActiGraph GT3X+ Accelerometer.
  Arms: Medium pace walking group

SUMMARY:
In this study, it will be investigated whether a daily 30-minute walk or abdominal breathing exercise is more effective on chronic constipation.

DETAILED DESCRIPTION:
According to the results of population-based studies conducted in our country, the frequency of constipation varies between 22-40%. In addition to medical treatment, alternative treatments are frequently used in the treatment of constipation. One of these is exercise.

In addition to medical treatment, alternative treatments are frequently used in the treatment of constipation. One of these is exercise. Many traditional breathing techniques developed in Asia are thought to be beneficial to health. In the light of this information, it is aimed to monitor ActiGraph GT3X+ Accelerometer, which is an objective measurement method of physical activity, and to evaluate the effectiveness of breathing exercise, which is one of the abdominal breathing exercises.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and understand Turkish,
* Voluntarily accepted to participate in the research and written consent form was obtained (those who could fill out the forms themselves using their hands, and those who could not use it, from their relatives with verbal consent),
* At least 18 years of age and over,
* Oriented to place, person and time,
* Patients who do not have spinal cord injury, parapilegia, or quadriplegia that may physiologically impede the individual's intestinal excretion Does not have any problems that prevent cognitive, sensory and verbal communication,
* Patients who are conscious and not using any sedating medication
* men and women aged 20-80 at the time of approval

Exclusion Criteria:

* pregnancy or possible pregnancy;
* the habit of doing all kinds of breathing exercises;

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | two months
  In order to determine the severity of constipation and the degree of impact of their current situation on their lives, individuals will be asked to mark a suitable point on a horizontal line with an actual length of 10 cm. In terms of the impact of the current situation on my life, "0" means it has no impact on my life, and "10" means living like this is unbearable.

SECONDARY OUTCOMES:
Constipation Severity Scale (CSS) | two months
  Constipation Severity Scale (CSS):There are 16 questions in total. The Constipation Severity Scale has three subscales: Fecal obstruction (FO), Large Intestinal Laziness (LIL) and Pain. The score that can be obtained from the FO sub-dimension is 0-28, the score that can be obtained from the LIL sub-dimension is 0-29,the score that can be received from the Pain sub-dimension is 0-16, and the lowest score that can be obtained from the CSS is 0 and the highest score is 73.High taken from the scale score indicates that symptoms are severe

OTHER OUTCOMES:
Chronic Constipation Quality of Life Scale | two months
  The PAC-QOL survey consists of 28 questions, and based on the factor analysis structure, the instrument consists of four subscales: "Physical discomfort (questions 1-4)," "Psychosocial discomfort (questions 5-12)," "Worries and concerns." (questions 13-23)" and "Satisfaction (questions 24-28)." Similar to a Likert scale, each option is scored from 0-4 (least to greatest impact), with higher scores indicating the worst quality of life. However, since questions 18, 25, 26, 27 and 28 were positive and the other 23 questions were negative, reverse coding was required.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Erdeo, Ph D, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Faculty of Nezahat Keleşoğlu Health Sciences Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No